CLINICAL TRIAL: NCT01081587
Title: Developing an Organization to Improve the Screening and Care of Starved Children in Hospital
Brief Title: Preventing Malnutrition and Restoring Nutritional Status in Hospitalized Children
Acronym: PREDIRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2008.522/23
Record Dates: First submitted 2010-02-19; First posted 2010-03-05 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Nutrition Disorders
Keywords: Non MeSH terms:; Children; Malnutrition; Computer Clinical Decision Support System; Cluster randomized trial; Healthcare workers; Guideline adherence; Patient safety; MeSH terms:; Nutrition Surveys; Secondary Prevention; Pediatrics; Child Care; Health Personnel; Reminder Systems; Intervention Studies; Quality of Health Care
MeSH Terms: conditions — Nutrition Disorders; Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nutritional Support Team (Experimental)
  Interventions: Procedure: Access to a Computerized Clinical Decision Support System (CCDDS); Behavioral: Education of Healthcare workers; Other: Local assistance by a dietician
- Usual care (Active Comparator)
  Interventions: Procedure: Access to a Computerized Clinical Decision Support System (CCDDS)

INTERVENTIONS:
Procedure: Access to a Computerized Clinical Decision Support System (CCDDS) — Automatic CCDSS will alert physician for each case of malnourished using an algorithm based on age, sex, weight and size of each hospitalized children.
Behavioral: Education of Healthcare workers — Education of the hospital staff to evidence-based practices in malnutrition care will be proposed in the experimental arm. Specific training will be targeted on participants according to their function.
  Arms: Nutritional Support Team
Other: Local assistance by a dietician — Assistance will be conducted locally by a local dietician. Periodic multidisciplinary meetings will be attended by the hospital staff belonging to the intervention arm, including the analysis of clinical incidents related to nutrition care.
  Arms: Nutritional Support Team

SUMMARY:
This cluster-randomized trial will evaluate the impact of a multifaceted intervention (including electronic medical alerts) coordinated by a Nutritional Support Team, on adherence to recommended practices for care of starved children, among health personnel of a large university hospital. A key component of the study is to assess whether improved adherence to guidelines leads to a reduction in rates of complications.

ELIGIBILITY:
Inclusion Criteria:

* medical and surgical units in a large teaching hospital providing pediatric acute care.
* any hospital staff with direct patient care who are affiliated with a single unit (includes physicians, nurses, nursing assistants, physiotherapists, dieticians.
* all children recorded as malnourished at their entrance in hospital

Exclusion Criteria:

* neonatal and intensive care units.
* any hospital staff with direct patient care who are not affiliated with a single unit.
* age under one month, liver or kidney abnormalities, severe heart failure, stay less than 2 days.

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1457 (Actual)
Dates: Start 2009-10; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Adherence to recommended practices (including weigh in, physiotherapy, nutrition survey and monitoring) | At least 2 days depending on the hospitalisation time

SECONDARY OUTCOMES:
Incidence of complications | At least 2 days depending on the hospitalisation time
Nutritional status evolution | At least 2 days depending on the hospitalisation time
Mean length and cost of stay | At least 2 days depending on the hospitalisation time
Appropriate call-in Nutritional Support Team | At least 2 days depending on the hospitalisation time

CONTACTS AND LOCATIONS:
Overall Officials: Noël PERETTI, MD, PhD, Principal Investigator — Hospices Civils de Lyon, Hôpital Femme-Mère-Enfant (Bron, France)
Locations (1):
- Hospices Civils de Lyon (HCL) - Hôpital Femme-Mère-Enfant, Bron, France

REFERENCES:
- [Result] Touzet S, Duclos A, Denis A, Restier-Miron L, Occelli P, Polazzi S, Betito D, Gamba G, Cour-Andlauer F, Colin C, Lachaux A, Peretti N; PREDIRE Study Group. Multifaceted intervention to enhance the screening and care of hospitalised malnourished children: study protocol for the PREDIRE cluster randomized controlled trial. BMC Health Serv Res. 2013 Mar 22;13:107. doi: 10.1186/1472-6963-13-107. PMID 23517767
- [Result] Duclos A, Touzet S, Restier L, Occelli P, Cour-Andlauer F, Denis A, Polazzi S, Colin C, Lachaux A, Peretti N; PREDIRE Study Group. Implementation of a computerized system in pediatric wards to improve nutritional care: a cluster randomized trial. Eur J Clin Nutr. 2015 Jul;69(7):769-75. doi: 10.1038/ejcn.2014.288. Epub 2015 Feb 4. PMID 25649237